CLINICAL TRIAL: NCT06763952
Title: Leveraging Artificial Intelligence to Prevent Vision Loss From Diabetes Among Socioeconomically Disadvantaged Communities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-0030; Version 8/9/24 (Other: UW Madison); A536000 (Other: UW Madison); 1R01EY035994 (NIH)
Record Dates: First submitted 2024-12-26; First posted 2025-01-08 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Vision; Diabetes
Keywords: Artificial Intelligence; AI; diabetic eye disease; cluster randomized trial; pragmatic trial
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: A stepped-wedge cluster randomized clinical trial will be conducted to evaluate the effectiveness of two standard diabetic retinopathy screenings across 9 underserved primary care clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care Screening (No Intervention): Primary care providers refer patients with diabetes to an eye care provider for a dilated eye exam. Patients are provided with culturally adapted diabetic eye disease educational materials similar to that provided to patients in the AI-BRIDGE group.
- AI-BRIDGE (Experimental): AI-based eye screening program called AI-Based point of caRe, Incorporating Diagnosis, SchedulinG, and Education (AI-BRIDGE). Eye photos of the patients will be obtained in the primary care clinic during a patient's regular primary care visit by a trained technician. Images will be reviewed using autonomous artificial-intelligence (AI) algorithm (Digital Diagnostics). Patients with referrable diabetic retinopathy are detected, and assisted with scheduling an in-person follow-up eye care visits. All patients irrespective of diabetic retinopathy status are also provided culturally adapted educational material on diabetic eye disease.
  Interventions: Other: AI-BRIDGE

INTERVENTIONS:
Other: AI-BRIDGE — AI-based eye screening program
  Arms: AI-BRIDGE

SUMMARY:
This study aims to investigate whether a novel artificial intelligence based screening strategy (AI-Based point of caRe, Incorporating Diagnosis, SchedulinG, and Education or AI-BRIDGE), which allows primary care providers to screen patients for vision-threatening diabetic eye disease in the primary care clinic, improves screening and follow-up care rates across race/ethnicity groups and reduces racial/ethnic disparities in screening.

DETAILED DESCRIPTION:
This is a multicenter clinical trial and University of Wisconsin is the coordinating center of the study.

A stepped-wedge cluster randomized clinical trial will be conducted. The investigators will evaluate the effectiveness of two standard diabetic retinopathy screening strategies at primary care clinics; (1) AI-based eye screening program called AI-BRIDGE, eye photos of the patients will be obtained in the primary care clinic by trained clinic staff. Images will be reviewed using autonomous artificial-intelligence (AI) algorithm (Digital Diagnostics). Patients with referrable diabetic retinopathy are detected within minutes and patients with referrable disease will be assisted with scheduling an in-person follow-up eye care visit (2) usual care screening, primary care providers refer patients with diabetes to an eye care provider for an in-person dilated eye exam.

After adapting AI-BRIDGE protocols to clinics and training of clinic personnel, stepped wedge randomized clinical trial begins with sites transitioning from usual-care to AI-BRIDGE in 4 steps.

Primary Objective:

* Compare the proportion of patients, by race and ethnicity, who follow-up with recommended eye care in the AI-BRIDGE and usual-care arms within 6 months of the recommendation.

Secondary Objectives:

* Compare the difference in proportion of White vs Hispanic and White vs Black patients who get screening in the AI-BRIDGE and usual-care arms within 6 months of the recommendation.
* Compare proportion of patients, by race and ethnicity, who receive eye screening in the AI-BRIDGE and usual-care arms within 6 months of the recommendation.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients include patients older than 21 years
* Diagnosed with type 1 or 2 diabetes
* No known diabetic eye disease
* Medicaid as their primary insurance
* Not had an eye exam in the prior year

Exclusion Criteria:

-

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Who Follow Up With Recommended Eye Care | up to 6 months
  Proportion of patients, by race and ethnicity, who follow-up with recommended eye care in the AI-BRIDGE and usual-care arms within 6 months of the recommendation.

SECONDARY OUTCOMES:
Difference in Proportion of White vs Hispanic and White vs Black Participants Who Get Eye Screening | up to 6 months
  Difference in proportion of White vs Hispanic and White vs Black patients who get AI-BRIDGE and usual-care screening within 6 months of the recommendation.
Proportion of Participants By Race and Ethnicity Who Get Eye Screening | up to 6 months
  Proportion of Participants by race and ethnicity who get eye screening in the AI-BRIDGE and usual-care arms within 6 months of the recommendation.

OTHER OUTCOMES:
Level of Diabetic Retinopathy | up to 6 months
  The rate of diabetic retinopathy, count of unique diabetic retinopathy diagnosis divided by count of all enrolled patients, stratified by intervention, intervention and race and ethnicity groups, and intervention, race and ethnicity group, and clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Roomasa Channa, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes